CLINICAL TRIAL: NCT04330508
Title: Effects of Direct-acting Antiviral Agents on Cognitive Function, and Depression in Chronic Hepatitis C
Brief Title: Effects of Direct-acting Antiviral Agents on HCV Cognitive Function, and Depression in HCV Related Cirrhosis: A Prospective Clinical Trial
Status: Completed | Type: Observational
Sponsor: Post Graduate Institute of Medical Education and Research, Chandigarh (Other)
Responsible Party: Principal Investigator, Madhumita Premkumar, Assistant professor, Department of heaptology, Post Graduate Institute of Medical Education and Research, Chandigarh
Other Study IDs: IEC-D3/2018-866
Record Dates: First submitted 2020-03-23; First posted 2020-04-01 (Actual); Last update posted 2024-02-13 (Actual); Status verified 2024-02

CONDITIONS: Depression in Chronic Hepatitis C
Keywords: Neurocognition, Minimal hepatic encephalopathy, Direct antivirals, DAAs, Chronic hepatitis C
MeSH Terms: conditions — Hepatitis C, Chronic | interventions — Neuropsychological Tests

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Group A: Chronic hepatitis C without Cirrhosis
  Interventions: Other: Depression and Cognitive Tests
- Chronic hepatitis C with Cirrhosis
  Interventions: Other: Depression and Cognitive Tests
- Healthy Volunteers

INTERVENTIONS:
Other: Depression and Cognitive Tests — Health Related Quality of Life, neurocognitive tests, PHES
  Other Names: SF36
  Groups: Chronic hepatitis C with Cirrhosis; Group A

SUMMARY:
Minimal hepatic encephalopathy (MHE) is an important clinical variant of hepatic encephalopathy (HE), which occurs in up to 60-70% of patients with cirrhosis. The condition comprises a cognitive impairment, observed in patients with cirrhosis who have no clinical evidence of overt hepatic encephalopathy (OHE). It is associated with an increased incidence of road traffic accidents, reduced quality of life and it affects the ability to perform tasks of daily living. Successful treatment of hepatitis C has been reported to be associated with 62-84% reduction in all-cause mortality (deaths), 68-79% reduction in risk of HCC and 90% reduction in risk of liver transplantation. In addition, studies have shown that viral eradication may improve cognition when given interferon based regimens for HCV. With the available of safe, efficacious, all oral regimens for HCV, we plan to prospectively analyse the change in mood, depression and cognitive function in response to DAA therapy, in relation to outcomes of treatment.

DETAILED DESCRIPTION:
Investigations will be performed according to the Declaration of Helsinki and approval of the enrolment as well as the usage of patient blood samples for research purpose will be obtained from the institutional ethics committee, and written informed consent will be obtained from all patients.The primary analysis upon which the sample size consideration was based involved the comparison of the SVR subgroup and the subgroup of patients without SVR. For the sample size calculation, we a two-factorial design (time course × SVR) with the use of a two-way analysis of variance (ANOVA) analysis, a significance level of 5% and a statistical power of at least 80% to detect a medium effect size (d = 0.5) and thus to show a significant group difference. Based on this background, the optimal sample size is calculated to be a total of 102 subjects. To consider asymmetric subgroups and to allow for a moderate dropout rate and additional calculations (secondary study objectives), we aim to include a total of at least 150 study participants in each group with 25 healthy volunteers as controls.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-65 years and chronic HCV infection.
* Group A: Patients with hepatitis C (Non-cirrhotic) [n= 150]
* Group B: Patients with hepatitis C related compensated-cirrhosis [n= 150]
* Group C: Healthy volunteers [n= 25]

Exclusion Criteria:

* Current overt hepatic encephalopathy or during the last 1 month
* TIPS (transjugular intra- hepatic porto-systemic shunt)
* elective surgery planned within the next 8 weeks
* unable to give informed consent
* HIV infection
* chronic respiratory insufficiency
* current infection and receiving antibiotics
* renal failure (serum creatinine ≥ 1.5 mg/l)
* hepatocellular carcinoma,
* patient with other neurological disease
* intake of sedatives, antidepressants, benzodiazepines, or benzodiazepines-antagonists (flumazenil, neuromuscular blocking agents)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with Chronic hepatitis C Infection
Sampling Method: Non-Probability Sample
Enrollment: 385 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2021-10-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Cognitive performance | Day 0
  Computerized battery (Reaction times, simple and choice, visual memory, Number connection test, and Inhibitory Control Test)
Cognitive performance | 90 days after treatment completion
  Computerized battery (Reaction times, simple and choice, visual memory, Number connection test, and Inhibitory Control Test)
Cognitive performance using conventional tests | Day 0
  Psychometric hepatic encephalopathy score (PHES), Indian Version.
Cognitive performance using conventional tests | 90 days after treatment completion
  Psychometric hepatic encephalopathy score (PHES), Indian Version.
HRQOL by SF-36 | Day 0
HRQOL by SF-36 | 90 days after treatment completion

SECONDARY OUTCOMES:
Depression Scale | Day 0
  Beck's Depression Inventory (BDI) Generalized anxiety disorder (GAD 7 score) Psychometric hepatic encephalopathy Score (PHES) Montreal Cognitive assessment Score (MoCA Score)
Depression Scale | 90 days after treatment completion
  Beck's Depression Inventory (BDI) Generalized anxiety disorder (GAD 7 score) Psychometric hepatic encephalopathy Score (PHES) Montreal Cognitive assessment Score (MoCA Score)

CONTACTS AND LOCATIONS:
Overall Officials: Madhumita Premkumar, DM, Principal Investigator — Post Graduate Institute of Medical Education and Research, Chandigarh
Locations (1):
- Postgraduate Institute of Medical Education and Research, Chandigarh, India

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Butterworth RF. Editorial: rifaximin and minimal hepatic encephalopathy. Am J Gastroenterol. 2011 Feb;106(2):317-8. doi: 10.1038/ajg.2010.460. PMID 21301455
- [Background] Poordad FF. Review article: the burden of hepatic encephalopathy. Aliment Pharmacol Ther. 2007 Feb;25 Suppl 1:3-9. doi: 10.1111/j.1746-6342.2006.03215.x. PMID 17295846
- [Background] Amodio P, Montagnese S, Gatta A, Morgan MY. Characteristics of minimal hepatic encephalopathy. Metab Brain Dis. 2004 Dec;19(3-4):253-67. doi: 10.1023/b:mebr.0000043975.01841.de. PMID 15554421
- [Background] Kircheis G, Knoche A, Hilger N, Manhart F, Schnitzler A, Schulze H, Haussinger D. Hepatic encephalopathy and fitness to drive. Gastroenterology. 2009 Nov;137(5):1706-15.e1-9. doi: 10.1053/j.gastro.2009.08.003. Epub 2009 Aug 15. PMID 19686744
- [Background] Ortiz M, Cordoba J, Jacas C, Flavia M, Esteban R, Guardia J. Neuropsychological abnormalities in cirrhosis include learning impairment. J Hepatol. 2006 Jan;44(1):104-10. doi: 10.1016/j.jhep.2005.06.013. Epub 2005 Jul 11. PMID 16169117
- [Background] Bajaj JS, Schubert CM, Heuman DM, Wade JB, Gibson DP, Topaz A, Saeian K, Hafeezullah M, Bell DE, Sterling RK, Stravitz RT, Luketic V, White MB, Sanyal AJ. Persistence of cognitive impairment after resolution of overt hepatic encephalopathy. Gastroenterology. 2010 Jun;138(7):2332-40. doi: 10.1053/j.gastro.2010.02.015. Epub 2010 Feb 20. PMID 20178797
- [Background] Bajaj JS, Saeian K, Schubert CM, Hafeezullah M, Franco J, Varma RR, Gibson DP, Hoffmann RG, Stravitz RT, Heuman DM, Sterling RK, Shiffman M, Topaz A, Boyett S, Bell D, Sanyal AJ. Minimal hepatic encephalopathy is associated with motor vehicle crashes: the reality beyond the driving test. Hepatology. 2009 Oct;50(4):1175-83. doi: 10.1002/hep.23128. PMID 19670416
- [Background] Conn HO. Trailmaking and number-connection tests in the assessment of mental state in portal systemic encephalopathy. Am J Dig Dis. 1977 Jun;22(6):541-50. doi: 10.1007/BF01072510. No abstract available. PMID 868833
- [Derived] Kaur H, Dhiman RK, Kulkarni AV, Premkumar M, Singh V, Duseja AK, Grover S, Grover GS, Roy A, Verma N, De A, Taneja S, Mehtani R, Mishra S, Kaur H. Improvement of chronic HCV infection-related depression, anxiety, and neurocognitive performance in persons achieving SVR-12: A real-world cohort study. J Viral Hepat. 2022 May;29(5):395-406. doi: 10.1111/jvh.13668. Epub 2022 Mar 17. PMID 35266624